CLINICAL TRIAL: NCT01770522
Title: A Longitudinal Study Exploring Factors Influencing Weight Gain During Pregnancy and Subsequent Weight Loss and Retention up to One Year Postpartum
Brief Title: Managing Weight in Pregnancy
Acronym: MAGIC
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 12068
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Pregnancy Related
Keywords: Bodyweight; Physical Acivitiy; Diet; Bodymass index; Pregnancy; Postnatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
It is well known that being overweight or obese increases the risk of health problems, and that many people find it difficult to maintain a healthy weight. Worryingly the rise in obesity is greater in women than in the male population. One possible reason for this is that some women gain too much weight during their pregnancy and find it difficult to lose this weight after the birth of their baby. For example, women who gain more weight than recommended during pregnancy have been shown to be more likely to carry excess that weight at 1 and 15 years after pregnancy, compared to women who gained the recommended amount of weight.

There are currently no evidence-based guidelines in the UK for how weight should be managed during pregnancy. For these reasons, it is really important that we understand the factors affecting weight management before, during and after pregnancy.

The aim of this research is therefore to find successful approaches to help women manage their weight before, during and after pregnancy. This will be completed by understanding the knowledge, attitudes, experiences and expectations of women during and after pregnancy and to identify the factors (e.g. diet, physical activity, poor social network etc.) which influence body weight. This will enable us to suggest better strategies for promoting healthy weight changes during and after pregnancy.

DETAILED DESCRIPTION:
Obesity in women of reproductive age is a major factor facing primary and secondary healthcare provision, with half of women of childbearing age in the UK classified as overweight or obese (The Information Centre, 2008). The prevalence of obesity in pregnant women living in Nottingham City is estimated to be 18.4%, (Wilcox, 2011), compared to 15.5% in England as a whole (Heslehurst et al., 2010). Being overweight or obese during pregnancy increases the risk of morbidity and mortality attributed to a range of pregnancy-related complications (Galtier et al, 2008), with 49% of maternal deaths occurring in overweight or obese women (Cantwell et al., 2011). Women who are overweight or obese at conception are more likely to develop hypertensive or diabetic complications, to develop thrombosis, and to deliver macrosomic babies (Ramachenderan et al, 2008). Associated with this are increased rates of delivery complications, postpartum haemorrhage and caesarean section (Galtier et al., 2008), with obese women at greater risk of anaesthetic complications. There is also a greater risk of infections (Metwally et al, 2007). Risks posed to the baby include congenital abnormalities such as spina bifida and oral clefts (King, 2006), and an increased risk of childhood obesity and adult metabolic syndrome (Galtier et al, 2008). The societal and economic impact of obesity during pregnancy is therefore life-long.

Excessive weight gain during pregnancy has little positive effect on foetal growth and pregnancy duration (Scholl et al, 1995) and is associated with a similar range of adverse outcomes as described above (Guelinckx et al., 2008). It is also associated with a greater probability of post-partum weight retention. Linné et al (2004) showed that both normal weight and overweight/obese women who gained excessive weight were more likely to have retained more weight 1 and 15 years after pregnancy, compared to women who gained the recommended amount of weight during pregnancy.

Whilst the US Institute of Medicine recommends lower pregnancy weight gain ranges for overweight and obese women (IOM, 2009), there are currently no UK evidence based guidelines outlining an appropriate BMI-specific weight gain (NICE, 2009). The current UK guide for weight gain is 10 - 12.5kg for all women (DoH, 2009). There is concern expressed that women are not being informed of the risks associated with obesity during pregnancy, or of the importance of a safe weight gain during pregnancy (NICE, 2009).

A study on the views of health professionals highlighted the issue that dietary information is often ad-hoc, and that advice is not linked with weight management (Heslehurst et al, 2007). Wiles (1998) found that above average weight women felt they didn't receive relevant weight management information. NICE (2010) recommended that there was need for research to find effective and cost effective approaches to help women manage their weight before, during and after pregnancy, including those from disadvantaged, low income and minority ethnic groups. In order to develop better strategies for promoting healthy weight changes in this population, it is important to understand the knowledge, attitudes and beliefs, experience and expectations of pregnant women during and after pregnancy in relation to their body weight and the behavioural factors which influence body weight. However, there is a paucity of research in this field. A recent systematic review (Campbell, et al, 2008) identified just 8 studies, (in the UK since 1990, with the most recent being conducted in 2004), into the views and attitudes to diet, physical activity and weight gain in pregnancy.

Childbearing may affect attitudes towards body image and this psychological dimension of weight is also important in understanding postpartum weight retention. Relatively few studies have investigated the effects of risk factors on weight retention in postpartum women. Gaining this intelligence from representative population groups is necessary for the selection and development of effective strategies to aid the development and commissioning of services and pathways to help address maternal obesity and post partum weight management.

Aim The primary risk factor for retaining weight in the postnatal period is excessive gestational weight gain (Linne et al., 2002). However, a number of other factors have been associated with an increased risk of weight retention, including high pre-pregnancy body mass index (BMI), primiparity, short duration of breastfeeding, stopping smoking, high dietary energy intake and low physical activity (Gunderson et al., 2000; Gore et al., 2003; Siega-Riz et al., 2004). Childbearing may also affect attitudes towards body image and this psychological dimension is important in understanding postnatal weight management. Understanding the effects of these risk factors on antenatal weight management is challenging and relatively few studies have attempted investigation of these relationships. Much of the data is inconclusive or focused on the effect of weight loss on other endpoints, such as lactation or infant growth (Dewey et al., 1994; Lovelady et al., 2000). Thus, the principal research objective of this project is to conduct a feasibility study to explore women's expectations and experiences of antenatal weight management and retention, and to use this to identify predictors of excessive weight gain during pregnancy and weight retention up to one year postpartum. Women will be recruited from antenatal clinics at Queens Medical Centre (Nottingham University Hospitals, NG7 2UH) at either 12 or 20 weeks of pregnancy. Parameters of interest will be investigated at recruitment whilst attending the antenatal clinic (12 or 20 weeks of pregnancy), at follow up during pregnancy by postal questionnaire (20 and 32 weeks of pregnancy), and at follow up during the postnatal period (2 weeks, 6 and 12 months after birth). The questionnaires will assess women's expectations for weight change during and after pregnancy, their experiences of antenatal care and knowledge of recommendations, and their diet and levels of physical activity. The participants will be women of all ages, sociodemographic backgrounds and bodyweights.

PURPOSE Purpose: The study has a clear purpose to explore women's expectations and experiences of antenatal weight management and retention, and to identify predictors of excessive weight gain during pregnancy and weight retention up to one year postpartum. It is imperative that these research questions are addressed in order to provide the knowledge required to develop appropriate intervention strategies. This study has been designed to address these research questions in a direct and focused manner, by using a combination of tools to collect the relevant information (questionnaire to explore women's expectations and experiences, food frequency and physical activity questionnaires). The ultimate aim is that the data collected will be used to develop intervention strategies to help women reach and/or maintain a healthy weight during the pregnancy and postnatal periods, thus reducing the risk of postpartum obesity.

PRIMARY OBJECTIVE The principal research objective is to conduct an exploratory, observational, mixed-methods study to assess women's expectations for weight change during and after pregnancy, their experiences of antenatal care and knowledge of recommendations, and their diet and levels of physical activity, and to use this information to identify predictors of weight change during pregnancy and the postnatal period that could usefully be targeted as part of an intervention.

SECONDARY OBJECTIVES

1. To determine what expectations women have with regards to weight change during pregnancy and the postpartum period.
2. To explore the sources of information which shape the expectations of women in relation to pregnancy-related weight change.
3. To determine whether the following factors are associated with weight change in pregnancy:

   1. Pre-pregnancy weight and body mass index.
   2. Diet and dietary habits during pregnancy.
   3. Physical activity during pregnancy.
   4. Pregnancy related symptoms.
4. To explore whether the following physiological factors predict weight change in post-partum women:

   1. Pre-pregnancy weight, pregnancy weight change and postpartum weight
   2. Diet and dietary habits during pregnancy and postpartum
   3. Physical activity during pregnancy and postpartum
   4. Breastfeeding, mixed or formula feeding, time of weaning
5. To identify whether the following psychological factors result in weight retention in post-partum women:

   1. Weight expectations
   2. Body weight and shape concerns
   3. Weight loss self-efficacy
   4. Body satisfaction
   5. Weight loss outcome expectancies

ELIGIBILITY:
Inclusion Criteria:

* Participants will be pregnant women at 12 or 20 weeks pregnancy attending the 12 and 20 week antenatal scanning clinics at the Queens Medical Centre, Nottingham
* Participants will be able to give informed consent- Participants will be over the age of 18
* Participants will be able to read English - due to the nature of the study we will not be able to print the questionnaires in various languages.
* Participants will be of any sociodemographic backgrounds, bodyweights and parity.

Exclusion Criteria:

* Participants who do not feel that their literacy or English language skills will enable them to complete the questionnaires will be offered the opportunity to have one of the research team read the questions and fill in the answers for them. Whilst doing this and being sensitive to literacy and language issues, the nature of this feasibility study means that the research team will not offer an interpreting service or produce documents in languages other than English.
* Participants will be excluded from the postnatal phase of the study if they deliver their baby prematurely (before 37 weeks of gestation) or do not give birth to a live baby. These exclusions are required, as premature birth or fetal loss/still birth would be expected to have an impact on psychological and physiological aspects linked to weight management which are not relevant to our specific research objectives. Information on birth outcome will be gained by accessing hospital records, and only women who have given birth to a live baby after 37 weeks of gestation will be contacted by the study team in the postnatal period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Particpants will be approached at their routine 12 or 20 weeks prnatal scan at the antenatal scanning clinics at the Queens Medical Centre, Nottingham.
Sampling Method: Probability Sample
Enrollment: 368 (Actual)
Dates: Start 2013-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Weight change during pregnancy and postnatal period | 18 months +/- 2 months
  To determine the weight change during pregnancy and postnatal period related to pre-pregnancy weight

SECONDARY OUTCOMES:
Secondary outcomes | 18 months +/- 2 months
  Expectations for weight change during and after pregnancy, their experiences of antenatal care and knowledge of recommendations, and their diet and levels of physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Preeti H Jethwa, PhD, Principal Investigator — University of Nottingham; Helen Budge, PhD, Principal Investigator — Queens Medical Centre
Locations (1):
- Univeristy of Nottingham Hospital, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Currently there is no plan to share data with other researchers, only publications

REFERENCES:
- [Background] Swift JA, Pearce J, Jethwa PH, Taylor MA, Avery A, Ellis S, Langley-Evans SC, McMullen S. Antenatal Weight Management: Women's Experiences, Behaviours, and Expectations of Weighing in Early Pregnancy. J Pregnancy. 2016;2016:8454759. doi: 10.1155/2016/8454759. Epub 2016 Oct 24. PMID 27843648
- [Result] Swift JA, Langley-Evans SC, Pearce J, Jethwa PH, Taylor MA, Avery A, Ellis S, McMullen S, Elliott-Sale KJ. Antenatal weight management: Diet, physical activity, and gestational weight gain in early pregnancy. Midwifery. 2017 Jun;49:40-46. doi: 10.1016/j.midw.2017.01.016. Epub 2017 Jan 31. PMID 28238351